CLINICAL TRIAL: NCT06942130
Title: Model Construction for AI-assisted Teaching
Brief Title: The Application of Artificial Intelligence in Dental Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital of Stomatology, Wuhan University (Other)
Responsible Party: Principal Investigator, Siyu Huang, MSM, Hospital of Stomatology, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024ZG147
Record Dates: First submitted 2025-04-14; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Medical Education
MeSH Terms: interventions — Artificial Intelligence; Videotape Recording

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial intelligence-assisted learning group (Experimental): After completing theoretical knowledge learning, students can use artificial intelligence for skills learning. AI provides steps for specific skill operations, points to note, as well as the desired performance and potential consequences of the operations.
  Interventions: Other: Artificial intelligence; Other: Video
- Control group (Active Comparator): This group is provided with detailed videos of specific clinical procedures, recorded by experienced physicians and educators, which demonstrate proper techniques and expected outcomes.
  Interventions: Other: Video

INTERVENTIONS:
Other: Artificial intelligence — Incorporating artificial intelligence as an aid to video-based skill learning
  Arms: Artificial intelligence-assisted learning group
Other: Video — Skill learning solely through videos

SUMMARY:
Clinical procedural skills training is a cornerstone of preclinical education for dental students. While technological aids such as virtual reality and simulators are increasingly integrated into training, direct instructor guidance remains fundamental to skill development. Artificial intelligence（AI）， as an emerging technology, is now gradually being adopted in medical education. This medical education trial, aimed at evaluating the potential of artificial intelligence in dental education, seeks to address two key questions: 1) Can AI assistance enhance the skill performance of dental students? 2) How can AI be effectively integrated into modern medical education? Researchers will compare the effects of AI and video-based instruction on skill acquisition, assessing differences in skill performance outcomes. Participants will engage in skill acquisition using either AI or video-based instruction over a one-week period.

ELIGIBILITY:
Inclusion Criteria:

* They must have completed courses in endodontics, periodontology, prosthodontics, and oral and maxillofacial surgery; participants should have little to no prior training in the skills related to the experiment; and they must voluntarily agree to participate in the study and sign an informed consent form.

Exclusion Criteria:

* Participants will be excluded if they meet any of the following criteria: failure in final exams of the four courses (endodontics, periodontology, prosthodontics, and oral and maxillofacial surgery); transfer to another major, suspension, or withdrawal from the current academic year; refusal to join the study or withdrawal midway; failure to meet the calibration standards in the 9-point eye-tracking calibration; use of OpenAI-related software or applications in the control group; or failure to complete the skill test.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Operational test scores | through study completion, an average 1 week
  Operational testing is a common method used to measure participants' proficiency in skill operation. At the conclusion of the experiment, participants completed a 15-minute operational test in a desktop VR environment. Scores were automatically calculated by the VR system, ensuring objectivity in the results.
spatial ability | Baseline
  Spatial ability, also known as visual-spatial ability (VSA) encompasses critical cognitive functions that enable individuals to understand, interpret, and manipulate spatially related information. The Purdue Spatial Visualization Test: Rotations (PSVT: R) - served as the measurement tool for analyzing subjects' mental rotation skills. This standardized evaluation contains 30 items that measure how effectively individuals can manipulate imagined three-dimensional figures. Each question includes an example and five choices, with only one being correct. Participants were tasked to rotate the given figure mentally in a similar manner as it was rotated in the example and to select the appropriate choice.
cognitive load | through study completion, an average 1 week
  Cognitive load refers to the resources required by working memory for a particular task. Eye-tracking technology has gained increasing popularity in investigating learners' visual attention distribution and cognitive load. As one of the key indicators, pupil diameter has been used to measure cognitive load during learning. In this study, we used eye-tracking devices to record the pupil diameter of participants during learning to quantify cognitive load.

SECONDARY OUTCOMES:
learning motivation | through study completion, an average 1 week
  Motivation is a motivational tendency guiding and sustaining a student's learning behavior toward specific academic goals.This study employed questionnaires to measure it. The questionnaire contains five items focusing on the motivation domain . Each item was coded according to a five-point Likert rating scale (1 = "strongly disagree", 2 = "disagree", 3 = "neutral", 4 = "agree", 5 = "strongly agree").
self-efficacy | through study completion, an average 1 week
  Self-efficacy, a concept first developed by Bandura, refers to people's subjective judgments regarding their ability to successfully perform an achievement behavior. The questionnaire contains five items focusing on the motivation domain . Each item was coded according to a five-point Likert rating scale (1 = "strongly disagree", 2 = "disagree", 3 = "neutral", 4 = "agree", 5 = "strongly agree").

CONTACTS AND LOCATIONS:
Overall Officials: Yang Dong, PhD, Study Chair — State Key Laboratory of Oral & Maxillofacial Reconstruction and Regeneration, Key Laboratory of Oral Biomedicine Ministry of Education, Hubei Key Laboratory of Stomatology, School & Hospital of Stomatology, Wuhan University
Locations (1):
- School & Hospital of Stomatology, Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang S, Wen C, Bai X, Li S, Wang S, Wang X, Yang D. Exploring the Application Capability of ChatGPT as an Instructor in Skills Education for Dental Medical Students: Randomized Controlled Trial. J Med Internet Res. 2025 May 27;27:e68538. doi: 10.2196/68538. PMID 40424023